CLINICAL TRIAL: NCT01920256
Title: Provider-Initiated Regular Remote Interventions for Optimal Type 2 Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Israel Hodish MD PhD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMichigan
Record Dates: First submitted 2013-08-02; First posted 2013-08-09 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes
Keywords: Insulin therapy; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized type 2 diabetes care. (Experimental): Remote, personalized type 2 diabetes clinic provided by an endocrinologist using frequent remote contacts for medication adjustments.
  Interventions: Other: Remote, personalized type 2 diabetes care.
- Usual Endocrine Care (Active Comparator): Usual Endocrine care will be provided by an endocrinologist.
  Interventions: Other: Usual Endocrine care.

INTERVENTIONS:
Other: Remote, personalized type 2 diabetes care. — Diabetes and comorbidities will be managed with 1 clinic visit per year and frequent adjustments made remotely.
  Arms: Personalized type 2 diabetes care.
Other: Usual Endocrine care. — Diabetes and comorbidities management will provided by an endocrinologist
  Arms: Usual Endocrine Care

SUMMARY:
Patients with type 2 diabetes can attain superior disease outcomes if multiple therapy goals are simultaneously achieved and maintained. In reality, therapy goals are seldom achieved, and patients become susceptible to devastating complications and greater health care expenses. Studies have shown that regular monitoring and therapy adjustments are a prerequisite to achieving and maintaining therapy goals. Unfortunately implementation of regular monitoring and therapy adjustments have been hindered by high clinic workload and shortage of endocrinologists. Due to this shortage, endocrine care is accessible to less than 20% of patients with type 2 diabetes. The overwhelming majority are managed by providers who may lack the necessary expertise or time to deliver optimal disease management, particularly when insulin is prescribed.

Objectives: We hypothesize that type 2 diabetes endocrine clinics for high-risk patients that complement primary care, personalize the frequency of remote disease interventions and employ infrequent face-to-face outpatient visits, will achieve comparable clinical outcomes and patient satisfaction compared to usual endocrine clinic care, while reducing workload and increasing the clinic capacity. The intervention clinic will employ regular remote communications initiated by the endocrinologists, based on tailored individual plans. Frequent remote monitoring and interventions will reinforce attainment of the therapy goals and allow a decrease in the frequency of outpatient visits. In turn, the clinic workload will decrease and it will be able to accommodate more patients with type 2 diabetes than traditional endocrine clinics. The aims of the study are to test this new endocrine clinic model in a clinical trial by monitoring clinical parameters, patient satisfaction and clinical workload. The long-term objectives are to modify the current model of endocrine care for patients with type 2 diabetes.

DETAILED DESCRIPTION:
Emerging data suggests that clinical interventions may be implemented successfully by a variety of remote communications. Thus far regular monitoring and treatment adjustments by remote communications have not yet been fully integrated into endocrine practice in a scalable fashion that can be readily disseminated. The PI proposes to test a new endocrine model care clinic for high-risk patients with type 2 diabetes that employs regular communications initiated by the provider, based on a tailored individual plan. Frequent monitoring and interventions will reinforce attainment of prespecified therapy goals, enhance patient engagement, and allow a significant decrease in the frequency of outpatient visits. In turn, the clinic will be able to accommodate more patients with type 2 diabetes than traditional endocrine clinics. Data management and day-to-day clinic operation will be computerized with technology that has been developed by the institution. The project is highly significant since it proposes a new model of endocrine care for high-risk patients with type 2 diabetes that may improved disease outcome in more patients and reduce medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years of age;
* Clinical diagnosis of type 2 diabetes (as defined by the American Diabetes Association 2);
* Treated with insulin or at least two diabetes medications;
* Have A1C ≥8.0% and ≤11.0%;
* Able and willing to use telephone or other sorts of communication regularly between clinic visits.

Exclusion Criteria:

* Do not speak English;
* Unwilling or unable to provide informed consent;
* Have any condition associated with life expectancy of less than 3 years;
* Have an active mental illness or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in baseline A1C (glycated hemoglobin) at 12 months | 12 months
  Measure of long-term blood glucose control and efficacy of intervention

SECONDARY OUTCOMES:
Change in baseline lipids at 12 months | 12 months
  Measure of total cholesterol, LDL, and Triglycerides
Change in baseline blood pressure at 12 months | 12 months
  Systolic and diastolic blood pressure
All cause mortality | 12 months
  Record deaths due to any cause
Acute complications | 12 months
  Cardiovascular events, cerebrovascular events, peripheral vascular events, limb ulcers and amputations, severe hypoglycemia, and other unscheduled emergency department and hospital visits
Change in baseline Quality of life at 12 months | 12 months
  Short Form-36
Change in baseline insulin satisfaction at 12 months | 12 months
  Insulin Therapy Satisfaction Questionnaire

OTHER OUTCOMES:
Clinic retention | 12 months
  Missed visits, missed phone calls, lost to follow up and drops outs will be recorded for both groups
Cost | 12 months
  Resource utilization and cost for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Israel Hodish, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Experimental group patients informed of A1C results.

REFERENCES:
- [Background] Klingeman H, Funnell M, Jhand A, Lathkar-Pradhan S, Hodish I. Type 2 diabetes specialty clinic model for the accountable care organization era. J Diabetes Complications. 2017 Oct;31(10):1521-1526. doi: 10.1016/j.jdiacomp.2017.05.011. Epub 2017 May 25. PMID 28793967